- 1 The effect of high intensity interval training and surgical weight loss on distal symmetric
- 2 polyneuropathy outcomes.
- 3 **July 2, 2025**

9

- 4 Statistical analysis
- 5 Our primary analysis was to determine the effect of HIIT and bariatric surgery on change in
- 6 IENFD of the proximal thigh during follow-up compared to the control group. Thus, the primary
- 7 covariate of interest was the interaction effect between follow-up time and treatment group.
- 8 Analysis of other outcomes was considered secondary analysis.
- Descriptive statistics were used to summarize participant demographic information at baseline.
- Within participant change was reported for metabolic phenotyping and neuropathy outcomes.
- For continuous variables, change was determined by subtracting baseline values from those at 2
- year follow up visit. For categorical variables, change was determined as those that improved
- from baseline to 2 year follow up visit. Paired t tests were used to compare within-participant
- change for continuous variables and the Wilcoxon signed rank test was used to compare within-
- participant change for ordinal categorical variables. Welch two sample t-tests (for continuous
- variables) and Persons's chi-squared tests (for categorical variables) were used to compare the
- within-participant change between each treatment and the no treatment group.
- 19 To account for non-compliance bias, the overall exercise compliance proportion was calculated
- 20 by adding the total compliant visits between baseline and the 2 year follow up visit and dividing
- 21 it by the total number of expected compliant visits in this period among those in HIIT

- 1 intervention group. Time varying compliance proportions specific to each follow up visit was
- 2 also calculated in a similar way by only considering the HIIT sessions occurring within each
- 3 follow up window. Compliance proportion was categorized into three groups: less than half a
- 4 session HIIT per week, less than one HIIT session per week and one or more HIIT session per
- 5 week. Compliance was assigned as zero for those not in HIIT intervention group.
- 6 Linear, poisson and zero inflation poisson mixed models were fitted to determine the effect of
- 7 each treatment with time on neuropathy outcomes. Since patients were not randomized to receive
- 8 surgery, we predicted the odds of receiving surgery using demographics and all models were
- 9 adjusted for this exposure. In addition, IENDF models were also adjusted separately for
- 10 circumferences at the biopsy locations. Sensitivity analysis was carried out to account for the
- effect of exercise compliance on neuropathy outcomes. We carried out a couple of different
- approaches: 1. Linear regression models to assess the association between treatment and within-
- participant change in outcomes between baseline and 2-year visit. Exercise was modelled using
- compliance proportions. 2. Linear, poisson and zero inflation poisson mixed models were rerun
- separately using exercise compliance proportions as numerical and categorical variables. A two
- tailed p-value with a cut-off of 0.05 was used to indicate statistical significance. All analyses
- were completed using R version (4.4.3)